CLINICAL TRIAL: NCT03088176
Title: A Phase 1b Trial of Talimogene Laherparepvec in Combination With Dabrafenib and Trametinib in Advanced Melanoma With an Activating BRAF Mutation
Brief Title: Combining Talimogene Laherparepvec With BRAF and MEK Inhibitors in BRAF Mutated Advanced Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: West Cancer Center (Other)
Collaborators: University of Tennessee (Other); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCC20149189
Record Dates: First submitted 2017-03-07; First posted 2017-03-23 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Melanoma; BRAF Gene Mutation
Keywords: Melanoma; BRAF inhibitor; Intratumoral injection; Talimogene laherparepvec; MEK inhibitor; dabrafenib; trametinib
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Phase 1b single arm single dose level
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination (Experimental): Talimogene laherperepvec intratumoral injection up to 4ml of 10^6 PFU/mL on Day 1, followed by up to 4mL of 10^8 PFU/mL 3 weeks later, followed by every 2 weeks thereafter for up to two years.
  Dabrafenib 150mg orally twice daily for up to two years Trametinib 2mg orally once daily for up to two years
  Interventions: Drug: Talimogene Laherparepvec 1 Million Pfu/Ml Inj,Susp,1Ml,Vil; Drug: Talimogene Laherparep 100 Mil Pfu/Ml 1Ml; Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Talimogene Laherparepvec 1 Million Pfu/Ml Inj,Susp,1Ml,Vil — Up to 4mL administered on C1D1 intratumorally
  Other Names: Imlygic
Drug: Talimogene Laherparep 100 Mil Pfu/Ml 1Ml — Up to 4 ML administered on Week 4 Day 1 and every 2 weeks thereafter
  Other Names: Imlygic
Drug: Dabrafenib — 150mg PO qday
  Other Names: Tafinlar
Drug: Trametinib — 2mg PO qday
  Other Names: Mekinist

SUMMARY:
The purpose of the study is to determine safety and tolerability of the combination of talimogene laherparepvec in combination with dabrafenib and trametinib in BRAF mutated advanced melanoma.

DETAILED DESCRIPTION:
While targeted therapies can successfully block oncogenic signaling in BRAF mutant melanoma, activation of an immune response with agents such as talimogene laherparepvec can induce durable responses in a subset of patients. Combining BRAF inhibitors and immunotherapy may specifically target the BRAF driver mutation in the tumor cells and potentially sensitize the immune system to target tumors.

The study will enroll up to 20 patients with advanced melanoma and activating mutations in the BRAF gene for the local administration of talimogene laherparepvec in conjunction with oral therapy with dabrafenib and trametinib, to describe the safety and tolerability of this combination.

Talimogene laherparepvec will be administered by intralesional injection into injectable cutaneous, subcutaneous, or nodal lesions with or without image ultrasound guidance. Talimogene laherparepvec will not be administered into any visceral organ or mucosal membrane lesions. The initial dose of talimogene laherparepvec is up to 4.0 mL of 106 plaque forming units (PFU)/mL. Subsequent doses of talimogene laherparepvec are up to 4.0 mL of 108 PFU/mL. The second dose of talimogene laherparepvec (the first dose of the 108 PFU formulation), will be administered at least 21 days following the initial dose. Subsequent doses will be given approximately every 2 weeks.

Dabrafenib at a dose of 150mg will be self-administered orally twice per day. Trametinib at a dose 2mg will be self-administered orally once per day.

Subjects will be evaluated by physical exam at the beginning of Cycle 1 (Week 1), Cycle 2 (Week 4), Cycle 3 (Week 6), Cycle 4 (Week 8), and every two cycles thereafter. Subjects will be evaluated for dose-limiting toxicities (defined in protocol) at Cycle 2 (Week 4), Cycle 3 (Week 6), and Cycle 4 (Week 8). Efficacy evaluation will be performed by tumor measurements using clinical assessment, CT or PET/CT every 4 cycles with the first non-baseline measurement prior to Cycle 4. Tumor response will be evaluated using RECIST 1.1. Adverse events will be recorded and graded using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0). Other safety assessments will include clinical laboratory values and physical exam findings. Reporting of adverse events, serious adverse events, and documentation of concomitant medications will occur as needed and at every cycle. Biopsy of a melanoma lesion (preferably uninjected) should occur at least one day prior to Cycle 4 (Week 8). Blood for biomarker analysis will be obtained immediately prior to the on-treatment biopsy, or if the on-treatment biopsy cannot be performed, immediately prior to Cycle 4 (Week 8).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Primary or recurrent Stage IIIB to IVM1c melanoma for whom surgery is not recommended
3. Activating BRAF mutation (limited to V600E or V600K mutations if being treated first-line, but can include any well-defined BRAF mutation after failure of prior immunotherapy)
4. Measurable disease defined as follows: At least one melanoma lesion that can be accurately and serially measured in one dimension and for which the longest diameter is ≥10 mm as measured by calipers, CT scan, or MRI.

   a. If all lesions are lymph nodes, at least one node must be able to be accurately and serially measured in two dimensions, and the short-axis must be ≥15mm.
5. Injectable disease (defined as at least 1cm of disease in areas suitable for injection including cutaneous, subcutaneous, or nodal lesions)

Exclusion Criteria:

1. Prior therapy with talimogene laherparepvec
2. Prior therapy with the combination of dabrafenib and trametinib
3. Evidence of clinically significant immunosuppression such as the following:

   1. Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
   2. Concurrent opportunistic infection
   3. Receiving chronic systemic immunosuppressive therapy (> 2 weeks), including oral steroid doses > 10mg/day of prednisone or equivalent except for management of adverse events and CNS metastases during the course of the study. Subjects requiring intermittent use of bronchodilators or local steroid injections are not excluded.
4. Active herpes infection, herpes requiring chronic anti-herpetic therapy, or complications of prior herpetic infection (such as keratitis or encephalitis)
5. Chronic use of immunosuppressants or steroids (defined as prednisone 10mg/day or equivalent)
6. Clinically active cerebral metastases
7. History or evidence of melanoma associated with immunodeficiency states
8. History of other malignancy within prior 24 months with the exception of breast or bladder carcinoma in situ, and non-melanomatous skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Dose Limiting Toxicities (DLT) | 2 years
  Number of DLT seen in the subject population

SECONDARY OUTCOMES:
Progression Free Survival | 4 years
  per RECIST 1.1
Objective Response Rate | 4 years
  per RECIST 1.1
Change in tumor burden | 4 years
  Best change in tumor diameters
Time to Response | 4 years
  In responding patients, time from first dose to achieving objective response
Duration of Response | 4 years
  In responding patients, time from first evidence of objective response until progression or end of study

OTHER OUTCOMES:
Lesion-level objective response | 4 years
  Change in diameters of individual lesions
Biomarker analysis | 4 years
  Exploratory analysis including number of participants with changes in CD8+ tumor infiltrating lymphocytes between pre-study and on-study biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- West Cancer Center, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified before publication or sharing with external entities or researchers